CLINICAL TRIAL: NCT06209281
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase III Clinical Study of the Efficacy and Safety of Two Low-concentration Atropine Sulfate Eye Drops in Slowing the Progression of Myopia in Children
Brief Title: A Phase III Clinical Study of the Efficacy and Safety of Two Low-concentration Atropine Sulfate Eye Drops
Acronym: Mini-CHAMP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-ATP-202105-Mini-CHAMP
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Experimental): 1 drop each time, once every night at bedtime
  Interventions: Drug: Lower dose atropine sulfate eye drops; Drug: Low dose atropine sulfate eye drops
- Experimental group 2 (Experimental): 1 drop each time, once every night at bedtime
  Interventions: Drug: Low dose atropine sulfate eye drops
- control group (Experimental): 1 drop each time, once every night at bedtime
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lower dose atropine sulfate eye drops — Administer to eyes
  Other Names: Eye drops
  Arms: Experimental group 1
Drug: Low dose atropine sulfate eye drops — Administer to eyes
  Other Names: Eye drops
  Arms: Experimental group 1; Experimental group 2
Drug: placebo — Administer to eyes
  Other Names: Eye drops
  Arms: control group

SUMMARY:
This study was a randomized, double-blind, placebo-controlled, multicenter, superiority design, phase III clinical trial to compare the efficacy and safety of two low-concentration atropine sulfate eye drops versus placebo in delaying myopia progression in children.

DETAILED DESCRIPTION:
Eligible subjects were screened and randomly assigned to the placebo control group, the lower dose group, and the lower dose group. Subjects received the study drug in both eyes, 1 drop each time, once every night before sleep, for continuous administration.A total of 526 subjects were planned to be enrolled。

Statistical analyses were performed with the use of SAS software, version 9.4, without any specific description. All statistical tests were two-sided at a 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

1. Child (female or male) aged 6 to 10 years.
2. Myopia (SER of at least -0.50 D and no more myopic than -6.00 D) in each eye as measured by cycloplegic autorefraction.
3. If present, astigmatism of ≤1.50 D in each eye as measured by cycloplegic autorefraction.
4. Anisometropia SER of < 1.50 D as measured by cycloplegic autorefraction.

Exclusion Criteria:

1. History of any disease or syndrome that predisposed the subject to severe myopia (e.g.,Marfan syndrome, Stickler syndrome, retinopathy of prematurity).
2. History in either eye of abnormal ocular refractive anatomy (e.g., keratoconus, lenticonus,spherophakia).
3. Chronic use of any topical or systemic antimuscarinic/anticholinergic medications (e.g.,atropine, scopolamine, tropicamide) within 21 days prior to screening and/or anticipated need for chronic use during the study period (i.e., more than 7 consecutive days in 1 month or more than 30 total days in 1 year).

   Use of cycloplegic drops for dilated ocular exam was allowable.
4. Heart rate persistently (for more than 10 minutes) > 120 beats per minute.
5. Allergy to study drugs.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 526 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic Autorefraction(low) | twelve months
  Group difference in the proportion of subjects eyes with myopia progression (SER) less than -0.50 D at M12 visit with low atropine versus placebo.

SECONDARY OUTCOMES:
Cycloplegic Autorefraction(lower) | twelve months
  Group difference in the proportion of subjects eyes with myopia progression (SER) less than -0.50 D at M12 visit with lower atropine versus placebo.
Cycloplegic Autorefraction(SER) | twelve months
  Between-group difference in the mean change from baseline in SER at visit M12

OTHER OUTCOMES:
Axial Length | twelve months
  Between-group difference in the mean change from baseline in axial length at visit M12
Crystalline Lens Thickness | twelve months
  Between-group difference in the mean change from baseline in crystalline lens thickness at visit M12

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Qu, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No